CLINICAL TRIAL: NCT04439968
Title: Targeted Cerebral Saturations in Extremely Preterm Infants
Brief Title: Neonatal Brain Oxygenation Study
Acronym: BOX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Valerie Chock, M.D., M.S. Epi, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 56759
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Hypoxia
MeSH Terms: conditions — Hypoxia, Brain

STUDY DESIGN:
Intervention Model Description: randomized to 2 groups: Targeted NIRS monitoring vs Non-targeted, blinded NIRS monitoring
Who Masked: Outcomes Assessor
Masking Description: Assessors of neurodevelopmental outcome are blinded to targeted vs non-targeted monitoring
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Csats (Active Comparator): Subjects randomized to the targeted Csat arm will have NIRS monitoring of cerebral saturations (Csat) and will have algorithm-driven clinical interventions to maintain Csat within target range in the first week of life.
  Interventions: Other: Clinical algorithm
- Non-targeted Csats (No Intervention): Subjects randomized to the non-targeted Csat arm will have NIRS (near-infrared spectroscopy) monitoring of Csats, but Csat values will be obscured and not available to providers. These subjects will not have any algorithm-driven clinical interventions for Csat.

INTERVENTIONS:
Other: Clinical algorithm — In order to maintain cerebral saturations within targeted range, subjects in the targeted Csat arm will undergo clinical interventions based on clinical algorithm. Interventions may include administration of inotropes, fluid resuscitation, transfusion of blood products, and/or adjustment to respiratory support.
  Arms: Targeted Csats

SUMMARY:
Implementing target ranges for regional cerebral saturations in extremely preterm infants in the first week of life may improve neurodevelopmental outcomes at 22-26 months corrected age compared to those without targeted cerebral saturations (Csat) using near-infrared spectroscopy (NIRS). Infants will be randomized to a targeted cerebral saturation monitoring group with visible reading of Csat or to a control group with cerebral saturation monitoring, but with blinded Csat measures. Those in the targeted Csat group will follow a treatment guideline to maintain cerebral oxygenation in the target range. The primary outcome is neurodevelopmental outcome as determined by Bayley III cognitive scale score.

ELIGIBILITY:
Inclusion Criteria:

* Very preterm infants with gestational age at least 23 weeks but less than 29 completed weeks
* Less than 6 hours of age

Exclusion Criteria:

* Skin integrity insufficient to allow placement of NIRS sensors
* Decision not to provide full intensive care support
* Congenital condition, other than premature birth, that adversely affects life expectancy or neurodevelopment

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcome | 22-26 months of age
  Neurodevelopmental outcomes will be assessed using the cognitive component of the Bayley Scales of Infant Development-III at 22-26 months of age. Scores range from 55-145 with higher number representing a better neurodevelopmental outcome.

SECONDARY OUTCOMES:
Death | from birth until hospital discharge, an average of 3 months.
  Death prior to hospital discharge
Retinopathy of prematurity | from birth until hospital discharge, an average of 3 months.
  Occurrence of retinopathy of prematurity prior to hospital discharge

OTHER OUTCOMES:
Burden of Cerebral hypoxia or hyperoxia | From birth until first 7 days of life
  Burden of cerebral hypoxia or hyperoxia from NIRS measures

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided